CLINICAL TRIAL: NCT03458533
Title: Changes in the Hypothalamic-pituitary Region of Patients With Metabolic Syndrome and Obesity
Brief Title: Changes in the Hypotalamic-pituitary Region of Patients With Metabolic Syndrome and Obesity
Acronym: CHIASM
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Andrea M. Isidori, MD, PhD, University of Roma La Sapienza
Other Study IDs: 4249
Record Dates: First submitted 2018-03-01; First posted 2018-03-08 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Overweight and Obesity; Metabolic Syndrome
Keywords: Pituitary; Obesity; Overweight; Metabolic syndrome; MRI
MeSH Terms: conditions — Overweight; Obesity; Metabolic Syndrome; Pituitary Diseases | interventions — Bariatric Surgery; Gastric Bypass; Diet; Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Obese patients with indication to bariatric surgery
  Interventions: Procedure: Bariatric surgery
- Group 2: Overweight or obese patients without indication to bariatric surgery, able to obtain weight loss trough diet and lifestyle changes
  Interventions: Behavioral: Diet and lifestyle changes
- Group 3: Overweight or obese patients without indication to bariatric surgery, not able to obtain weight loss trough diet and lifestyle changes
  Interventions: Behavioral: Diet and lifestyle changes

INTERVENTIONS:
Procedure: Bariatric surgery
  Other Names: sleeve gastrectomy; gastric bypass; bilio-intestinal bypass
  Groups: Group 1
Behavioral: Diet and lifestyle changes
  Other Names: hypocaloric diet; physical exercise
  Groups: Group 2; Group 3

SUMMARY:
This study aims to identify new morphological and quantitative magnetic imaging parameters of pituitary gland and sellar region in overweight and obese patient at baseline and after 3 years, dividing patients in 3 groups (weight loss through diet and lifestyle changes, weight loss through bariatric surgery, no weight loss)

DETAILED DESCRIPTION:
This longitudinal prospective study in overweight and obese patients aims to identify and characterize new morphological and quantitative MRI parameters of pituitary gland and sellar region assessed by texture analysis with a specific software (ImageJ©). These parameters will be correlated them to hypothalamic-pituitary-peripheral axis function, metabolism and body composition.

Data will be detected at baseline and at 3 years follow-up to quantitatively identify the different pituitary MRI patterns in 3 groups:

1. patients without weight modifies
2. patients with weight loss obtain through diet and lifestyle changes
3. patients with weight loss obtained through bariatric surgery

ELIGIBILITY:
Inclusion Criteria:

* BMI > 25 Kg/m2

Exclusion Criteria:

* Malignant neoplasia;
* Current use of psychotropic drugs;
* Chronic renal failure;
* Pituitary macroadenomas and craniopharyngiomas;
* Contraindications to MRI execution (p. e. pace-maker, metal foreign bodies like slivers, non MRI compatible vascular clips or prosthesis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Overweight and obese patients come to our attention for weight loss interventions
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Pituitary volume | 0, +3 years
  Change in pituitary volume (mm3) from baseline to 3 years

SECONDARY OUTCOMES:
Evaluation of pituitary mean and standard deviation intensity | 0, +3 years
  Changes in new quantitative magnetic imaging parameters of pituitary gland from baseline to 3 years
Correlation of magnetic resonance parameters with anthropometric measurements | 0, +3 years
  Correlation analysis of pituitary mean and standard deviation intensity with anthropometric measurements
Correlation of magnetic resonance parameters with pituitary axis function | 0, +3 years
  Correlation analysis of pituitary mean and standard deviation intensity with pituitary axis function
Correlation of magnetic resonance parameters with glyco-metabolic status | 0, +3 years
  Correlation analysis of pituitary mean and standard deviation intensity with glyco-metabolic status

CONTACTS AND LOCATIONS:
Overall Officials: Andrea M Isidori, MD, PhD, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Andrea M Isidori, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Puliani G, Sbardella E, Cozzolino A, Sada V, Tozzi R, Andreoli C, Fiorelli M, Di Biasi C, Corallino D, Balla A, Paganini AM, Venneri MA, Lenzi A, Lubrano C, Isidori AM. Pituitary T1 signal intensity at magnetic resonance imaging is reduced in patients with obesity: results from the CHIASM study. Int J Obes (Lond). 2023 Oct;47(10):948-955. doi: 10.1038/s41366-023-01338-w. Epub 2023 Jul 21. PMID 37479795